CLINICAL TRIAL: NCT05638074
Title: Does the Presence of Cervical Facet Tropism Affect the Response to Interlaminar Epidural Steroid Injections? A Prospective Clinical Study
Brief Title: Does the Presence of Cervical Facet Tropism Affect the Response to Interlaminar Epidural Steroid Injections?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Janbubi Jandaulyet (Other)
Responsible Party: Sponsor-Investigator, Janbubi Jandaulyet, Resident Doctor, Marmara University
Organization: Marmara University (Other)
Other Study IDs: 04.11.2022.1506
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Cervical Disc Herniation; Cervical Radicular Pain; Facet Tropism
Keywords: facet tropism; cervical disc herniation; Cervical Radicular Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- With cervical facet tropism
  Interventions: Procedure: Interlaminar Epidural Steroid Injection
- Without cervical facet tropism
  Interventions: Procedure: Interlaminar Epidural Steroid Injection

INTERVENTIONS:
Procedure: Interlaminar Epidural Steroid Injection — The patient will be placed in the prone position and cutaneous anesthesia is performed with 3 mL of 2% prilocaine using the sterile technique. After imaging the C7-T1 space with fluoroscopy, it will be entered from the right/left paramedian part of the C7-T1 space with an 18G Touhy needle, and the C-arm will be set in the contralateral oblique position for depth determination.
  Under intermittent fluoroscopic imaging, the needle will be advanced, and access to the epidural space wiil be confirmed by the loss of resistance technique. Afterwards, the epidural spread will be controlled with a contrast agent, and a mixture of 10 mg dexamethasone, 1 mL 2% lidocaine hydrochloride, and 1 mL 0.9% saline will be applied to the epidural space. The patient will be discharged with recommendations after being kept under observation for 2 hours post-procedure. All injections will be performed by the same pain medicine specialist who has at least 5 years of experience.

SUMMARY:
Facet joints are synovial joints located on the dorsolateral side of the vertebral column. Normally, both facet joints are symmetrical. Facet tropism (FT) is defined as asymmetry between the angles of orientation of the joints, in which a facet joint in the same segment is more sagittally oriented than the other. In 1967, Farfan and Sullivan first reported that FT is a possible risk factor for the development of disk herniation. However, this is controversial as there are other views advocating that FT is not a risk factor for the development of cervical disc herniation. Further, it has been emphasized that patients with FT have a greater need for adjacent segment degeneration and new spinal surgery after spinal fusion surgeries than those without FT.

In the current literature, studies have been conducted to examine the clinical and radiological parameters that may be related to the effectiveness of cervical interlaminar epidural steroid injections (ILESI). The aim of this study was to examine the effect of the presence of FT on ILESI results in patients with cervical disc herniation-induced radicular pain.

ELIGIBILITY:
Inclusion Criteria:

aged 18-75 years, who applied to the pain medicine outpatient clinic, had axial neck and unilateral radicular extremity pain for at least 3 months, and were diagnosed with protruded disc herniation by magnetic resonance imaging were included in the study

Exclusion Criteria:

Patients with systemic inflammatory disease, bleeding diathesis,history of psychiatric illness, malignancy, contrast material or local anesthetic agent allergy, cervical spinal stenosis, history of cervical ESI, or neck surgery in the last 3 months were excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to the pain medicine outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-11-28 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
NRS score | at first hour, at three weeks, at 3 months
  ≥50% reduction in the NRS scores at month 3 relative to the initial NRS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Hakan Gunduz, Professor, Study Director — Marmara University
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Celenlioglu AE, Sencan S, Gunduz OH. Does facet tropism negatively affect the response to transforaminal epidural steroid injections? A prospective clinical study. Skeletal Radiol. 2019 Jul;48(7):1051-1058. doi: 10.1007/s00256-018-3129-8. Epub 2019 Jan 2. PMID 30603772